CLINICAL TRIAL: NCT06028399
Title: Effects of Concurrent Training on Glycaemic & Vascular Parameters Among Patients With Type-II DM Associated Peripheral Artery Disease.
Brief Title: Concurrent Training on Patients With Type-II DM Associated PAD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Uroosa Amin, Student, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7170523HSPAT
Record Dates: First submitted 2023-08-30; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes With Peripheral Angiopathy
Keywords: Concurrent Exercise Training; Physical Exercise; Glycated hemoglobin; Glycemic control; Insulin Resistance; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Motor Activity; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, there are 2 parallel groups. Group A for Concurrent training and Group B for Aerobic training.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be allocated to the intervention group by using sealed envelop methods of simple random sampling. They were masked for the treatment allocation group. For assessment of outcome measures, HbA1C will be assessed by lab investigator, ABI and Functioncal capacity will be assessed by the physiotherapist who will be supervised the session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Training (Experimental): Concurrent training combines aerobic and resistance training within the same session for 30 - 60 minutes, comprising 3 sessions per week for 12 weeks.
  Interventions: Other: Concurrent Training
- Aerobic Training (Active Comparator): Aerobic training for 30 - 60 minutes comprises 3 sessions per week for 12 weeks.
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Other: Concurrent Training — The patient in the Concurrent Training group will perform exercises for 30 - 60 minutes in 3 sessions per week for 12 weeks under the supervision of a physical therapist. Aerobic training will be performed on a treadmill at an intensity of 40 - 60 % THR for 15 - 40 minutes, followed by resistance training (Quadriceps extension, leg curls, calf raise & toe raise) using an elastic resistance band at an intensity of 60 - 80% of 1 RM, following appropriate rest intervals.
  Arms: Concurrent Training
Other: Aerobic Training — The patient in the Aerobic Training group will perform exercises on a treadmill for 30 - 60 minutes in 3 sessions per week for 12 weeks under the supervision of a physical therapist. Aerobic training will be performed on a treadmill at an intensity of 40 - 60 % THR, following appropriate rest intervals.
  Arms: Aerobic Training

SUMMARY:
This clinical trial aims to analyze the effects of concurrent vs aerobic training on glycemic control, ABI, functional capacity and disease-specific QOL among patients with Type-II DM-associated PAD at baseline & after 12 weeks of intervention. The main questions it aims to answer are:

1. Is concurrent training more effective than aerobic training in improving glycemic control among patients with Type-II DM-associated PAD?
2. Is concurrent training more effective than aerobic training in improving ABI among patients with Type-II DM-associated PAD?
3. Is concurrent training more effective than aerobic training in enhancing functional capacity among patients with Type-II DM-associated PAD?
4. Is concurrent training more effective than aerobic training in improving QOL among patients with Type-II DM-associated PAD? Signed informed consent will be taken before participation. For exercise training, Both will perform Warm up for 10 - 12 minutes, followed by 30 - 60 minutes of training protocol and then Cool down exercises for 10 - 12 minutes. Group A will perform concurrent training, whereas Group B will perform aerobic training.

DETAILED DESCRIPTION:
DATA COLLECTION PROCEDURE;

Eighty patients will be referred from the OPD of Dr. Ziauddin Hospital Karachi, Pakistan. Signed informed consent will be obtained before participation. In the screening session, PAD by Fontaine's stage IIa, ABI (<0.9), and an international Physical activity questionnaire (IPAQ) to assess sedentary behaviour will be collected. For IPAQ interpretation, <600 MET Minutes will be considered category 1 (Lowest level of physical activity). In the next session, baseline measurements of all participants will be collected and documented, including HbA1C, ABI at rest, Functional Capacity, and QOL.

Moreover, Target heart rate (THR) and 1RM will be calculated for appropriate exercise intensity and BMI. Further, All patients will be randomly allocated into two groups. Group A (n=40) will perform concurrent training, whereas Group B will perform aerobic training (n=40). All patients will receive a brief explanation and demonstration of the exercise session during the familiarisation. Patients will perform 3 sessions weekly to improve their capability to do exercises and develop the exercise capacity needed to begin at the intensity of their allocated training protocol. Both groups will perform warm-up exercises for 10 - 12 minutes during the training session, followed by training protocol and then cool-down exercises for 10 - 12 minutes. Group A will perform concurrent training for 30 to 60 minutes, whereas Group B will perform aerobic training for 30 - 60 minutes. Both groups will perform warm-up and cool-down exercises for 10 - 12 minutes, including 5 minutes of static cycling followed by 5 reps. of static stretching of the hamstring, quadriceps, and calf muscles on each limb with the 10-second hold of each stretch (ACSM, 2018). During the intervention period, patients will be assessed for Heart rate, blood pressure, and random blood sugar before and after each session for 12 weeks duration, and perceived exertion status will be used during exercise for analyzing the exercise intensity.

Group A (Concurrent Training):

Concurrent training combines aerobic and resistance training within the same session. Patients in this group will perform aerobic exercises and resistance training for 30 - 60 minutes, comprising 3 sessions per week for 12 weeks under the supervision of a physical therapist. Aerobic training will be performed on a treadmill at an intensity of 40 - 60 % THR for 15 - 40 minutes, followed by resistance training using an elastic resistance band at 60 - 80% of 1 RM, following appropriate rest intervals. The patient will perform lower limb resistance exercises, including Quadriceps extension, leg curls, calf raises & toe raises.

Group B (Aerobic Training):

Patients in this group will perform aerobic exercise for 12 weeks. All Patients will be assessed for HR, BP and RBS before and after each session. Patients in this group will perform aerobic exercises for 30 - 60 minutes, comprising 3 sessions per week for 12 weeks under the supervision of a physical therapist. Aerobic training will be performed on a treadmill at an intensity of 40 - 60 % THR.

After 12 weeks of intervention, all patients will be assessed for HbA1C, ABI, functional capacity, and QOL and documented for further data analysis.

SPECIAL CONSIDERATION FOR EXERCISE

* Educate the patient about the signs and symptoms of hypoglycemia.
* Hypoglycemia manifestations (particularly tachycardia) may mask due to Β-Blockers.
* Blood glucose level monitoring (before and after exercise).
* Carbohydrate intake (up to 15 g before exercise participation) to prevent hypoglycemia *when starting RBS ≤100 mg/dL.
* Avoid head-down activities and the Valsalva manoeuvre.
* For peripheral neuropathy, closely examine feet regularly to detect sores or ulcers and incorporate proper foot care (dry feet, silica gel or air midsoles & polyester socks).

EXERCISE TERMINATION CRITERIA The exercise will be terminated if the patient reports any following symptoms during exercise.

* The onset of Chest pain
* Shortness of breath (Borg's scale >15)
* Hemodynamic imbalance during exercise is caused by limited perfusion (Pale appearance, cool skin, Diaphoresis (sweating), Physical exertion, altered pulse) and Low blood pressure (very late sign)
* On the patient's request to stop exercise
* Ischemic limb pain that is not alleviated after 10 minutes

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 - 50 years
* Type-II DM
* Duration of DM: > 10 years
* Baseline HbA1C (> 6.6%)
* Intermittent claudication corresponding to Fontaine Stage IIa
* PAD by an ABI scale; < 0.9 at rest
* Had < 160 mmHg SBP and < 105 mmHg DBP
* Sedentary lifestyle by IPAQ-SF

Exclusion Criteria:

* Smokers
* Insulin dependent individuals
* Patients with Complicated cardiovascular disease that might limit their ability to - participate in the intervention period physically (e.g. unstable cardiopulmonary symptoms, ischemic heart failure, or chronic kidney disease) and cancer
* Any major surgery or revascularization procedure within the previous 1 year
* In case of a history of severe arthritis that may limit exercise performance
* Diabetic foot (ulceration or gangrene)
* Patients with stroke
* BMI = >30 classified by WHO-Asian as obesity class II
* Unable to follow the intervention protocol or visit three times per week for exercise
* Participation in any clinical trial during the past six months
* Revocation to consent

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
HbA1c for glycemic control | 12 weeks
  The hemoglobin A1C (HbA1c) is a gold standard for assessing glycemic control for 2-3 months (Chehregosha et al., 2019). HbA1C has excellent reliability and validity (Sn= 0.8, Sp=0.9, AUROC = 0.9) (Rathod et al., 2018).
Ankle Brachial Index (ABI) for peripheral artery disease | 12 weeks
  ABI is a non-invasive method for determining the presence and severity of PAD, commonly used in clinical settings (Thurston and Dawson, 2019). Doppler ABI has 80.3% sensitivity and 78.1% specificity on the side with high pressures (Mayr et al., 2019). An ABI of 0.9 is considered diagnostic for PAD. Using a portable Doppler Ultrasound with a 5MHz probe, the systolic pressures of the right and left brachial, & dorsalis pedis arteries will be assessed then higher systolic blood pressure will be considered for the study. The ABI will be calculated by dividing the brachial pressures by the lower extremity (Chen et al., 2021).
Functional Capacity for functional claudication distance | 12 weeks
  The patient will walk on 100 feet indoor track, and distance will be measured on claudication symptoms when the patient prefers to stop walking, which will analyze pre and post-intervention to assess the effectiveness of therapeutic intervention (Sinnige et al., 2022). The reliability of FCD is 0.959. FCD is a reliable and valid measurement for determining functional capacity in patients with intermittent claudication (Bubb et al., 2021, Abola et al., 2020).
Quality of life for disease-specific patient reported outcomes | 12 weeks
  The Vasculo-6 questionnaire evaluates disease-specific QOL among patients with symptomatic PAD. Each question is scored out of four, of which one is the lowest score, and four will be the highest. The sum of all components yields the final score. The final score could range between 6-24 points. VQ-6 has strong reliability (Cronbach=0.82), validity (AUC=0.754) & excellent receptivity to change after intervention (standard response means=1.12)

CONTACTS AND LOCATIONS:
Overall Officials: Uroosa Amin, DPT, Principal Investigator — Ziauddin University
Locations (1):
- Uroosa Amin, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No